CLINICAL TRIAL: NCT05237791
Title: Effect of Magnesium Sulfate on Remifentanil Induced Cough and Chest Wall Rigidity
Brief Title: Effect of Magnesium on Remifentanil Induced Cough
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B-2201-731-001
Record Dates: First submitted 2022-01-29; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium group (Experimental): magnesium sulphate 50mg/kg (loading dose for 10 minutes), 15mg/kg/hr (continuous infusion)
  Interventions: Drug: Magnesium sulfate
- control group (Placebo Comparator): normal saline 100ml (loading for 10 minutes), 15mg/kg/hr (continuous infusion)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium sulfate — magnesium sulphate 50mg/kg (loading dose for 10 minutes), 15mg/kg/hr (continuous infusion)
  Arms: magnesium group
Drug: Placebo — normal saline 100ml (loading dose for 10 minutes), 15mg/kg/hr (continuous infusion)
  Arms: control group

SUMMARY:
The hypothesis of this study is that Magnesium sulfate pretreatment (50mg/kg) will reduce the incidence of cough and chest wall rigidity caused by remifentanil administration.

The purpose of this study was to investigate the effect of magnesium sulfate administered before induction of anesthesia on thoracic stiffness and cough response caused by opioid analgesics administered for general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-75 years of age who are undergoing surgery under general anesthesia using a laryngeal mask and who have consented to participate in this study among American Society of Anesthesiologists body grade 1 or 2

Exclusion Criteria:

* When coughing may occur due to an underlying disease (upper respiratory infection, rhinitis, post nasal drip, asthma, chronic obstructive pulmonary disease, pneumonia, bronchitis, current smokers, etc.)
* If you have kidney disease that can affect magnesium metabolism (glomerular filtration rate less than 60)
* If you are taking opioid analgesics or magnesium for other reasons
* Patients with hypermagnesemia
* Patients with atrioventricular block (stages I-III) or other cardiac conduction disorders
* Pregnant or lactating women
* Patients with myasthenia gravis
* Patients taking drugs that are contraindicated or interact with magnesium (barbitalates, aminoglycoside antibiotics, isoniazid, chlorpromazine, digoxin)
* In case of hypersensitivity to magnesium
* Patients with a history of hypersensitivity to propofol and any of its components
* Patients with a history of hypersensitivity to remifentanil and other fentanyl analogues

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-02-03 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
remifentanil induced cough | from preoperative 20 minutes to induction of anesthesia
  To evaluate whether coughing occurs during anesthesia induction from the start of remifentanil infusion to the completion of laryngeal mask insertion.

SECONDARY OUTCOMES:
severity of cough | from preoperative 20 minutes to induction of anesthesia
  mild: 1-2, moderate: 3-4, severe: ≥ 5
laryngeal mask airway (LMA) insertion compliance | from preoperative 20 minutes to induction of anesthesia
  Assess the number of trials prior to successful laryngeal mask insertion and the need for administration of a neuromuscular blocker.
lung compliance | from induction of anesthesia to finish of surgery
  Poor compliance of mechanical ventilation is defined as a difference between the set tidal volume and the actual tidal volume value applied to the patient by 100ml or more.